CLINICAL TRIAL: NCT02768818
Title: Modulation of the Intestinal Flora With the Probiotic VIVOMIXX™ in Pregnant Women at Risk of Metabolic Complications
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Facchinetti Fabio, Chairman of Obstetrics and Gynecology Unit, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CE 91/14
Record Dates: First submitted 2016-04-20; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-01

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy, Diet- Controlled; Exercise Addiction; High-Risk Pregnancy; Dietary Modification
Keywords: Maternal Obesity Complicating Pregnancy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Intervention (Experimental): Probiotic VIVOMIXX™
  Interventions: Dietary Supplement: Probiotic VIVOMIXX™
- Control (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic VIVOMIXX™ — The patients will be randomly assigned to the VIVOMIXX™ (intervention) or the control (placebo) group through a randomization list elaborated by a specific software.
  Arms: Intervention
Dietary Supplement: Placebo — The patients will be randomly assigned to the VIVOMIXX™ (intervention) or the control (placebo) group through a randomization list elaborated by a specific software.
  Arms: Control

SUMMARY:
The investigators aimed at evaluating the effectiveness of probiotics ingestion in changing maternal microbiota and preventing gestational diabetes in overweight and obese women.

To achieve these goals, obese (BMI> 30 kg/m^2) or overweight (BMI> 25 kg/m^2) pregnant women with risk factors were enrolled in the study and randomized to the supplementation with the probiotic VIVOMIXX® or with placebo.

The endpoints of this study are to evaluate if the dietary supplementation with the probiotic VIVOMIXX® modifies the maternal fecal microbiota (bifidobacteria and lactobacilli) and related enzymatic activity (alkaline sphingomyelinase and alkaline phosphatase), and if this if this is linked to an improvement of the intermediate metabolism (positive Oral Glucose Tolerance Test at 24-26 weeks).

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled trial.

208 pregnant women from the recruiting centers will be enrolled as follow: Women eligible to participate, prior informed consent, will be randomized to 2 capsules twice daily before breakfast and before dinner from randomization until delivery. The boxes will be given to the patients coded and blinded to investigators and participants, and will contain either the active ingredient (VIVOMIXX®, a mixture of 112 billion of eight strains for each capsule, namely Streptococcus thermophilus, bifidobacteria (B. breve, B. longum, B. infantis) and lactobacilli (L. paracasei, L. acidophilus, L. delbrueckii subsp bulgaricus, L. plantarum) or placebo.

The protocol includes a screening visit (Visit 1) at 10-12 weeks, two visits during pregnancy (at 26-28 weeks= Visit 2, and at 36-38 weeks=Visit 3) and a postnatal visit (2-3 days after delivery=Visit 4).

Eligible women should take two capsules twice daily (2 in the morning and 2 in the evening). Patients will be randomly assigned to the control or the VIVOMIXX® group.

The study agent VIVOMIXX® as well as the placebo will be supplied by "Mendes SA" for the whole study period.

During Visit 1 (at 10-12 weeks) written consent will be obtained, after information on expected benefits and possible inconveniences related to participation in the trial. Furthermore, eligible women will be asked to complete two questionnaires, one on dietary habits and one on gastrointestinal symptoms. The questionnaire on gastrointestinal symptoms will be submitted to the patients at each visit.

Height will be assessed at Visit 1, while the following parameters will be measured at each visit: weight, waits/hip circumference ratio, arterial blood pressure, plasma hemoglobin (Hb), hematocrit (Ht), fasting glycemia, fasting insulin and fasting glycated hemoglobin (HbA1c1).

A blood sample for the evaluation of homocysteine will be taken as well as urine and a faeces sample will be collected for nuclear-magnetic-resonance (NMR)-based metabolomics and intestinal microbiota analysis.

Furthermore, an Arm-band will be positioned for monitoring sleep and physical activities for one week at each visit.

At Visit 2 and 3 data regarding ultrasound examinations (Amniotic fluid index, abdominal circumference, cephalic circumference ratio) will be also collected.

Two-three days after delivery (Visit 4) data regarding the delivery (mode of delivery, gestational age at delivery) as well as the newborn (Apgar score, glycemia and serum bilirubin) were collected.

Moreover, a sample of colostrum (for NMR-based metabolomics, microbiota and high performance liquid chromatography-mass spectrometry -HPLC/MS- of vitamins analysis) and newborn faeces (for NMR-based metabolomics and microbiota analysis) sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 40 with singleton pregnancies and BMI at recruitment > 30 kg/m^2 or a BMI> 25 kg/m^2 and the simultaneous presence of at least 1 of the following risk factors: age> 35 years, previous fetal macrosomia (> 4500gr), family history of diabetes (first-degree relative with type 2 diabetes mellitus), previous gestational diabetes mellitus.
* Adherence to lifestyle prescription including dietary counselling and physical activity stimulation

Exclusion Criteria:

* Subjects who require intervention in addition to the lifestyle changes women with diet and habits much different from the Mediterranean area (Central Africa, Asian, etc..). In such subgroup it will be difficult to obtain adherence to diet prescription since their cultural attitudes and dietary habits.
* Pre-pregnancy BMI> 40 kg/m^2
* Chronic hypertension
* Fasting glycemia in the first trimester of> 126 mg / dl or random glycemia > 200 mg/dl

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 205 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12

PRIMARY OUTCOMES:
Maternal and newborn fecal microbiota changes (bifidobacteria and lactobacilli) and related enzymatic activity (alkaline sphingomyelinase and alkaline phosphatase) modifications | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  NMR-based metabolomics, microbiota and high performance liquid chromatography-mass spectrometry -HPLC/MS- of vitamins analysis
Glucose metabolism changes | At 24-26 week
  Positive Oral Glucose Tolerance Test

SECONDARY OUTCOMES:
Weight changes | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  Measured in kg
Maternal BMI | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  Measured in kg/m^2
Waist/hip circumference ratio | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
Gestational weight gain | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  Measured in kg
HOMA Index | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
HbA1c1 | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
glycemia | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
insulinemia | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
homocysteine plasmatic levels | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
Requirement for insulin therapy | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  Week of onset
Requirement for insulin therapy | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  Dose of insulin
Quality of sleep | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  Hours of deep sleep measured through the armband
Duration of sleep | At baseline, at 24-26 week, at 36-38 week, 2-3 days after delivery
  Measured in hours through the armband
Onset of hypertension / preeclampsia | At delivery
Time of delivery | At delivery
Mode of delivery | At delivery
Complications during delivery | At delivery
  Surgery and/or hemorrhage >500ml and/or shoulder dystocia
Apgar score | Within 1 hour after delivery
Newborn's weight | Within 1 hour after delivery
Newborn's sex | Within 1 hour after delivery
Newborn's abdomen / head ratio | 2-3 days after delivery
Newborn's skinfold thickness at birth | 2-3 days after delivery
Neonatal hypoglycemia | Within 24 hours from delivery
  Neonatal hypoglycemia (measured in mg/dl) that requires therapy
Neonatal bilirubinemia | At delivery, 2-3 days after delivery
  Measured in mg/dl
Neonatal complications | 2-3 days after delivery
  Respiratory Distress Syndrome, Necrotizing Enterocolitis, Retinopathy of prematurity, Bronchopulmonary Dysplasia, Neonatal Death
Admission to Neonatal Intensive Care Unit (NICU) | Within 24 hours after delivery
  Admission to NICU
Admission to Neonatal Intensive Care Unit (NICU) | Within 24 hours after delivery
  Duration of stay at the NICU

CONTACTS AND LOCATIONS:
Locations (1):
- Mother-Infant Department, University of Modena and Reggio Emilia, Italy, Modena, Italy